CLINICAL TRIAL: NCT07122908
Title: The Effect of Repetitive Transcranial Magnetic Stimulation on Cognitive Improvement in Dementia With Lewy Bodies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Kyoungwon Baik, Clinical Assistant Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024AN0178
Record Dates: First submitted 2024-05-28; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 10Hz (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — 10Hz stimulation group will receive 1600 pulses of stimulation in a single session

SUMMARY:
This study aimed to investigate the feasibility of repetitive transcranial magnetic stimulation (rTMS) on the occipital lobe in patients with Lewy body dementia.

This is a proof-of-concept study to evaluate the safety and effect of occipital lobe stimulation in patients with Lewy body dementia. Over a period of two weeks, participants will receive rTMS to the primary visual cortex three times a week during visits. For the remaining 10 weeks, maintenance therapy will be administered with rTMS once a week during visits. Efficacy assessments will be conducted on the day of the final stimulation session and again four weeks later.

DETAILED DESCRIPTION:
This is a proof-of-concept, single-arm clinical study investigating the safety and potential cognitive benefits of repetitive transcranial magnetic stimulation (rTMS) in patients with dementia with Lewy bodies (DLB). All enrolled participants will receive active rTMS, delivered at 10 Hz over the primary visual cortex.

Following screening based on the 2017 criteria for probable DLB, eligible patients (aged ≥65 years, with a Clinical Dementia Rating [CDR] between 0.5 and 1.0) will undergo baseline EEG (Electroencephalography) and MRI (Magnetic resonance imaging) to exclude other causes of cognitive impairment. A single-pulse TMS session will be used to determine the phosphene threshold. rTMS sessions will then commence, with stimulation administered three times per week for 2 weeks (induction phase), followed by once-weekly sessions for 10 weeks (maintenance phase). Each rTMS session will deliver 1,600 pulses over 20 minutes (10 Hz frequency, 4-second trains with 26-second inter-train intervals).

Primary efficacy will be evaluated based on change in CDR-SOB (Clinical Dementia Rating - Sum of Boxes) from baseline to the end of treatment (week 12). Secondary outcomes include changes in MMSE (Mini-Mental State Examination), K-MOCA (Korean version of the Montreal Cognitive Assessment), CGA-NPI (Caregiver-Administered Neuropsychiatric Inventory), CGI (Clinical Global Impression), PGI (Patient's Global Impression). Assessments will be conducted at baseline, immediately after the last treatment session, and at a 4-week follow-up. Safety will be evaluated through adverse event monitoring, categorized by severity and relation to the intervention.

The intervention device is the Brain Hi ATNC-MDD V2 magnetic stimulator, used in conjunction with the ATNC-BN-V1 neuronavigation system. Devices will be managed by trained technicians throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years of age
* Meeting the criteria for Probable DLB as proposed in the 2017 DLB diagnostic criteria
* Scoring between 0.5 and 1 on the Clinical Dementia Rating Scale (CDR)

Exclusion Criteria:

* If other causes of cognitive impairment are suspected, such as neurosyphilis, hypothyroidism, hyperthyroidism, metabolic encephalopathy, brain tumor, acute cerebral hemorrhage, acute cerebral infarction, previous territorial or strategic cerebral infarction, Wernicke's encephalopathy, or severe white matter hyperintensity detected in hematological tests, brain MRI, etc.
* If cooperation for interviews and self-assessment is difficult (e.g., due to hearing impairment, language disorders, severe psychotic conditions)
* If there is a history of psychiatric disorders: major affective disorder, schizophrenia, or schizo-affective disorder
* If electroencephalography (EEG) cannot be performed
* If epileptiform EEG findings are present or if the patient is currently receiving antiepileptic drugs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sum of boxes of the clinical dementia rating scale | Week 12
  The Clinical Dementia Rating - Sum of Boxes (CDR-SOB) is a quantitative scale used to assess the severity of cognitive and functional impairment in individuals with dementia. It is derived from the Clinical Dementia Rating (CDR), which evaluates six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care.
  Each domain is rated on a scale from 0 (no impairment) to 3 (severe impairment), and the scores are summed to produce the CDR-SOB, which ranges from 0 to 18. Unlike the global CDR score, the CDR-SOB provides a more sensitive measure of changes in cognitive and functional performance over time, making it especially useful for tracking disease progression in clinical trials and longitudinal studies.

SECONDARY OUTCOMES:
Mini-Mental State Examination | Week 12
  A brief 30-point cognitive screening tool that assesses orientation, memory, attention, calculation, language, and visuospatial skills. 0-30 (higher = better cognition)
Korean version of the Montreal Cognitive Assessment | Week 12
  A more sensitive 30-point cognitive screening test than MMSE, used to detect mild cognitive impairment; assesses memory, executive function, attention, language, and visuospatial skills. 0-30 (higher = better cognition)
Caregiver-Administered Neuropsychiatric Inventory | Week 12
  A caregiver-based questionnaire evaluating behavioral and psychiatric symptoms in dementia across 12 domains (e.g., delusions, hallucinations, agitation). 0-144 (higher = worse symptoms; frequency × severity per domain)
Clinical Global Impression | Week 12
  Assessing overall treatment response. CGI-I: 1-7 (1 = very much improved, 7 = very much worse)
Patient's Global Impression | Week 12
  Patient's self-rating of their perception of change in overall health status after treatment. 1-7 (1 = very much improved, 7 = very much worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Due to regulation of institutional IRB